CLINICAL TRIAL: NCT06600932
Title: Effects of Transcranial Magnetic Stimulation on Visual Outcome in Patients After Cataract Surgery
Brief Title: Evaluation of TMS Visual Outcome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai High Myopia Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMSG2024015
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cataract Surgery Experience
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TMS (Experimental): TMS treatment indicates a non-invasive procedure called transcranial magnetic simulation (TMS) on cortex. The treatment intensity is set as 80% of the threshold of each participant. The treatment will be conducted every day for consecutive 5 days.
  Interventions: Procedure: TMS
- Control (Sham Comparator): The sham group will be exposed to the recorded sounds of TMS pulses but without real magnetic stimulation.
  Interventions: Procedure: control group

INTERVENTIONS:
Procedure: TMS — TMS treatment in this study indicates a non-invasive procedure called transcranial magnetic simulation (TMS) on visual cortex. The treatment intensity is set as 80% of the threshold of each participant. The treatment will be conducted every day for consecutive 5 days.
  Arms: TMS
Procedure: control group — The control treatment is a sham-controlled procedure, in which participants will be exposed to the recorded sounds of TMS pulses but without real magnetic stimulation.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if transcranial magnetic stimulation (TMS) can improve the visual outcomes in patients after cataract surgery. The main question it aims to answer is:

• Does TMS improve the visual outcome in patients after cataract surgery? Researchers will compare TMS to the sham-controlled treatment (exposure to recorded sounds of pulses without real magnetic stimulation) to see if TMS works to improve the visual outcomes of patients after cataract surgery.

Participants will

* Undergo TMS treatment or a sham-controlled treatment for consecutive 5 days.
* Visit the clinic once every 2 weeks for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* Post cataract surgery
* Best-corrected visual acuity less than 0.1logMAR

Exclusion Criteria:

* Diagnosed with cognitive impairment or mental disorders and unable to cooperate with treatment;
* Diagnosed with significant opacity of refractive media that affects observation of visual function;
* History of epileptic seizures;
* Long term use of psychotropic drugs；
* Metal implants in the body.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | From enrollment to the end of treatment at 2 weeks

SECONDARY OUTCOMES:
Visual field | From enrollment to the end of treatment at 2 weeks

OTHER OUTCOMES:
Visual quality | From enrollment to the end of treatment at 12 weeks
  Include objective visual quality (contrast sensitivity) and subjective visual quality (visual function questionnaire score).

CONTACTS AND LOCATIONS:
Overall Officials: Xiangjia Zhu, Study Chair — Eye and ENT Hospital of Fudan University; Jiaqi Meng, Principal Investigator — Eye and ENT Hospital of Fudan University; Yinglei Zhang, Principal Investigator — Eye and ENT Hospital of Fudan University; Yating Tang, Principal Investigator — Eye and ENT Hospital of Fudan University; Xin Liu, Principal Investigator — Eye and ENT Hospital of Fudan University
Locations (1):
- Eye and Ear, Nose Throat Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided